CLINICAL TRIAL: NCT04987502
Title: Virtual Reality and Subjective Tinnitus
Acronym: ReVA2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut de recherche et de coordination acoustique/musique (Unknown); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Immersive Therapy (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP210808; 2021-A01045-36 (Registry Identifier: ID-RCB Number - ANSM)
Record Dates: First submitted 2021-07-31; First posted 2021-08-03 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Tinnitus; Tinnitus, Subjective
Keywords: Subjective tinnitus; Virtual Reality; Cognitive Behavioral Therapy
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual reality treatment (Experimental): Virtual reality immersion with 3D audio and visual rendering (8 weekly sessions)
  Interventions: Other: Virtual Reality
- Standard treatment (Active Comparator): Counselling Relaxation techniques Sound enrichment
  Interventions: Behavioral: Standard treatment

INTERVENTIONS:
Other: Virtual Reality — 8 sessions of virtual reality with 3D audio and visual rendering
  Arms: Virtual reality treatment
Behavioral: Standard treatment — counselling, relaxation techniques, sound enrichment
  Arms: Standard treatment

SUMMARY:
The purpose of this study is to test if virtual reality immersion has the potential to significantly decrease subjective tinnitus intrusiveness when compared to standard care.

DETAILED DESCRIPTION:
This is a randomised controlled study aimed at further validating the use of Virtual Reality in the field of subjective tinnitus management. Indeed, earlier results have suggested that this innovative strategy has the potential to be as efficient as a Cognitive and Behavioural Therapy.

Before the sessions, an automated tinnitus matching procedure will help create a sound similar to the tinnitus percept ("Tinnitus Avatar").

During the sessions (8 sessions; 30 minutes), the "Tinnitus Avatar" will be displayed auditorily but also visually - as a sparkling spot - in a variety of virtual 3D auditory and visual environments.

In these virtual environments the patients will be given the possibility to voluntarily control and manipulate the "Tinnitus Avatar" by the means of a wand on top of which the sound and the sparkling will be attached. They will also be able to freely navigate in the virtual scenes where environmental sound will be displayed.

Then the patients will be able to displace at will the "Tinnitus Avatar" in their peri-personal space or mask it by getting close to sounds they may encounter in the virtual scenes.

It is supposed that regaining and training a capacity of interaction with the "Tinnitus Avatar" as if it were a standard sound will help recalibrate the attentional processes involved in tinnitus perception and then to decrease tinnitus intrusiveness.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years and < 75 years,
* French speaking and ability to understand multidimensional questionnaires,
* Subjective tinnitus of peripheral origin (middle or inner ear auditory nerve)
* Subjective tinnitus stable and chronic (lasting for more than 6 months)
* Subjective tinnitus that can be characterized by tinnitus matching
* Normal hearing or moderate hearing loss

Exclusion Criteria:

* Fluctuating tinnitus,
* Unilateral or bilateral severe or profound hearing loss,
* Claustrophobia, visual, impairment, vertigo or dizziness, chronic headache or any other condition contraindicating virtual immersion
* Psychiatric condition requiring immediate management
* Pregnant or breastfeeding women
* Protected adults (including individual under guardianship by court order)
* Persons deprived of their liberty by judicial or administrative decision

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Subjective Tinnitus Severity Scale (S.T.S.S.) | 5 months
  16 items multidimensional questionnaire (validated in French) Score 0 to 16 (maximum severity)

SECONDARY OUTCOMES:
Tinnitus Handicap Questionnaire (THI) | 5 months
  25 items multidimensional questionnaire (validated in French) Score 0 to 100 (maximum handicap)
Hospital Anxiety Depression Scale | 5 months
  14 item questionnaire (validated in French) Score 0 to 21 (maximum anxiety) Score 0 to 21 (maximum depression)
Visual Analog Scale Tinnitus Loudness | 5 months
  Likert-Scale 0 to 10 (maximum loudness)
Visual Analog Scale Tinnitus Intrusiveness | 5 months
  Likert-Scale 0 to 10 (maximum intrusiveness)

CONTACTS AND LOCATIONS:
Overall Officials: Alain Londero, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital européen Georges-Pompidou AP-HP, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered.
  Data sharing must respect the agreements made with funders. Teams wishing obtain IPD must meet the sponsor and IP team to present scientific (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractual agreement.
  Processing of shared data must comply with European General Data Protection Regulation (GDPR).

REFERENCES:
- [Background] Malinvaud D, Londero A, Niarra R, Peignard P, Warusfel O, Viaud-Delmon I, Chatellier G, Bonfils P. Auditory and visual 3D virtual reality therapy as a new treatment for chronic subjective tinnitus: Results of a randomized controlled trial. Hear Res. 2016 Mar;333:127-135. doi: 10.1016/j.heares.2015.12.023. Epub 2016 Jan 8. PMID 26773752